## STATISTICAL ANALYSIS PLAN

Title: A Double-Blind, Placebo-Controlled, Randomized, Multicenter, Proof of

Concept and Dose-Finding Phase II Clinical Trial to Investigate the Safety, Tolerability and Efficacy of ADRECIZUMAB in Patients with

Septic Shock and Elevated Adrenomedullin

Short Title: Treatment of patients with septic shock and bio-ADM concentration > 70

pg/mL with ADRECIZUMAB

Version / Date: Final 1.0 / 05-Feb-2020

Protocol No.: ADR-02

EudraCT-No: 2016-003883-38 NCT: NCT03085758

| | M.A.R.C.O. | Version: | 1.0 |
|-----|---------------------------|----------|--------------|
| _ | WI.7 (.1 (. C. C. | Date: | 05FEB2020 |
| - 1 | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## STATISTICAL ANALYSIS PLAN

# STUDY NUMBER: ADR-02 (ADRENOSS-2) CONFIDENTIAL

A Double-Blind, Placebo-Controlled, Randomized, Multicenter, Proof of Concept and Dose-Finding Phase II Clinical Trial to Investigate the Safety, Tolerability and Efficacy of ADRECIZUMAB in Patients with Septic Shock and Elevated Adrenomedullin

Sponsor: ADRENOMED AG

Neuendorfstr. 15a D-16761 Hennigsdorf

Germany

Author Jenni Reifenberger

M.A.R.C.O. GmbH & Co.KG

Schirmerstr. 71

D-40211 Duesseldorf

Phone: +49 (0)221/ 97793-579

Email: jenni.reifenberger@marco-institut.de

Version: 1.0

Date: 05<sup>th</sup> February 2020

#### **CONFIDENTIALITY STATEMENT**

The following confidential information is the property of ADRENOMED AG. All rights are strictly reserved. Reproductions of all or single sections of this protocol is not permitted. Acceptance of this document constitutes the agreement by the recipient that no unpublished information contained within will be published or disclosed to third parties without prior written approval, except that this document may be disclosed to the appropriate ethics committee and regulatory authority under the condition that they are requested to keep it confidential.

|---------------|---------------------------|-----------|--------------|
| IVI.A.IX.C.O. | Date: | 05FEB2020 | |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

| Dr. Jens Zimmermann, M.D., M.Sc.<br>Chief Medical Officer<br>ADRENOMED AG | Date |
|---|---|
| Dr. Oliver Hartmann<br>Senior Principal Statistician<br>ADRENOMED AG | Date |
| Jenni Reifenberger<br>Statistical Analyst<br>M.A.R.C.O. | Date |

## CONFIDENTIALITY STATEMENT

The following confidential information is the property of ADRENOMED AG. All rights are strictly reserved. Reproductions of all or single sections of this protocol is not permitted. Acceptance of this document constitutes the agreement by the recipient that no unpublished information contained within will be published or disclosed to third parties without prior written approval, except that this document may be disclosed to the appropriate ethics committee and regulatory authority under the condition that they are requested to keep it confidential.

|---------------------------|----------|--------------|
| <br>WI.71.11.0.0. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

Dr. Jens Zimmermann, M.D., M.Sc. Date Chief Medical Officer ADRENOMED AG

Dr. Oliver Hartmann Senior Principal Statistician ADRENOMED AG

Date

Jenni Reifenberger Date Statistical Analyst

M.A.R.C.O.

## CONFIDENTIALITY STATEMENT

The following confidential information is the property of ADRENOMED AG. All rights are strictly reserved. Reproductions of all or single sections of this protocol is not permitted. Acceptance of this document constitutes the agreement by the recipient that no unpublished information contained within will be published or disclosed to third parties without prior written approval, except that this document may be disclosed to the appropriate ethics committee and regulatory authority under the condition that they are requested to keep it confidential.

| | M.A.R.C.O. Statistical Analysis Plan | Version: | 1.0 |
|---|---|---|---|
| *************************************** | 141.71.11.0.0. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

Dr. Jens Zimmermann, M.D., M.Sc.

Chief Medical Officer ADRENOMED AG

05-FED-1010 Date

Dr. Oliver Hartmann Senior Principal Statistician ADRENOMED AG

Date

Jenni Reifenberger Date

M.A.R.C.O.

#### CONFIDENTIALITY STATEMENT

The following confidential information is the property of ADRENOMED AG. All rights are strictly reserved. Reproductions of all or single sections of this protocol is not permitted. Acceptance of this document constitutes the agreement by the recipient that no unpublished information contained within will be published or disclosed to third parties without prior written approval, except that this document may be disclosed to the appropriate ethics committee and regulatory authority under the condition that they are requested to keep it confidential.

|---|---------------------------|----------|------------------------|
| - | | Date: | 05FEB2020 |
| , | Statistical Analysis Plan | Project: | ADR-02<br>(AdrenOSS-2) |

Dr. Jens Zimmermann, M.D., M.Sc. Chief Medical Officer ADRENOMED AG

Date

Dr. Oliver Hartmann Senior Principal Statistician

ADRENOMED AG

Statistical Analyst

M.A.R.C.O.

05 FEB 2020

CONFIDENTIALITY STATEMENT

The following confidential information is the property of ADRENOMED AG. All rights are strictly reserved. Reproductions of all or single sections of this protocol is not permitted. Acceptance of this document constitutes the agreement by the recipient that no unpublished information contained within will be published or disclosed to third parties without prior written approval, except that this document may be disclosed to the appropriate ethics committee and regulatory authority under the condition that they are requested to keep it confidential.

## **Table of contents**

| LISTING | OF ABBREVIATIONS AND DEFINITION OF TERMS | 6 |
|---|---|---|
| 1. | BACKGROUND AND SCOPE | 8 |
| 2. | STUDY OBJECTIVES | 8 |
| 3. | STUDY DESIGN | 9 |
| 3.1. | Main characteristics of study design | 9 |
| 3.2. | Sample Size Determination / Power Analysis | 9 |
| 3.3. | Hypotheses | |
| 4. | PATIENT POPULATION | 10 |
| 5. | ENDPOINTS FOR PRIMARY AND SECONDARY OBJECTIVES AND EXPLORATORY ENDPOINTS | 11 |
| 5.1. | Endpoints for primary objectives | 11 |
| 5.2. | Endpoints for secondary objectives | 11 |
| 5.3. | Exploratory endpoints | |
| 6. | GENERAL CONVENTIONS | |
| 6.1. | Treatment groups | 12 |
| 6.2. | Layout of tables | 13 |
| 6.3. | General calculation rules | 14 |
| 6.4. | Descriptive statistics | 16 |
| 7. | ANALYSIS SETS AND DATA REVIEW CRITERIA | |
| 7.1. | Data sets for analysis | |
| 7.2. | Protocol violations/data review | 17 |
| 8. | DATA ANALYSIS | 18 |
| 8.1. | Statistical software | 18 |
| 8.2. | Definitions, derived variables and handling of missing data | |
| 8.2.1.<br>8.2.2. | Definitions of time points / time windows | |
| 8.2.3. | Derived variables Handling of missing values | |
| 8.3. | Sensitivity analyses | |
| 8.4. | Disposition | 26 |
| 8.5. | Demographic data and baseline characteristics | 27 |
| 8.6. | Analysis of primary endpoints | 28 |
| 8.7. | Analysis of secondary endpoints | 29 |
| 8.8. | Pharmacokinetic data analyses | 32 |

| M.A.R.C.O. | Version | 1.0 |
|---------------------------|----------|--------------|
| <br>WI.A.IX.C.O. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

| 8.8.1. | Pharmacokinetic parameters | 32 |
|---------|-----------------------------------------------|----|
| 8.8.2. | Analysis of pharmacokinetic endpoints | 33 |
| 8.8.3. | Descriptive pharmacokinetic analyses | 33 |
| 8.9. | Pharmacodynamic data analyses | 34 |
| 8.10. | Evaluation of relationships between endpoints | 34 |
| 8.11. | Safety analysis | 34 |
| 8.11.1. | Extent of exposure | |
| 8.11.2. | Adverse events | |
| 8.11.3. | Clinical laboratory | 35 |
| 8.11.4. | Vital signs and body temperature | |
| 8.11.5. | ECG | |
| 8.11.6. | Biomarker | |
| 8.11.7. | Other assessments | 36 |
| 9. | CHANGES TO THE PROTOCOL | 36 |
| 10. | CHANGES TO THE SAP AFTER FINALIZATION | 36 |
| 11. | CONTENTS OF STATISTICAL TABLES AND FIGURES | 37 |
| 12. | CONTENTS OF APPENDICES | 43 |
| 13. | DEFINITION OF SCORES | 44 |
| 13.1. | SOFA Score | 44 |
| 13.2. | APACHE II Score | |
| 14. | REFERENCES | 47 |

| | .A.R.C.O. | Version: | 1.0 |
|----------------|---------------------------|-----------|--------------|
| - WI.A.IV.C.O. | Date: | 05FEB2020 | |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## Listing of tables

| TABLE 1 | TREATMENT GROUPS AND SAMPLE SIZES | 9 |
|---------|-----------------------------------|----|
| TABLE 2 | LAYOUT OF TABLES1 | 13 |

|---------------------------|----------|--------------|
| - WI.A.IV.C.O. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

## Listing of abbreviations and definition of terms

ADM Adrenomedullin AE Adverse event

AUC Area under the curve

ATC Anatomic therapeutic class

Bio-ADM Biologically active Adrenomedullin, measured by Sphingotec bio-ADM assay

BLLOQ Below lower limit of quantification

BMI Body mass index

CCC Clinical Coordinating Center for central evaluation

CL Systemic clearance

C<sub>max</sub> Maximum concentration

CV Coefficient of variation

DPP3 Dipeptidyl-Peptidase 3

ECG Electrocardiogram

eCRF Electronic case report form

FAS Full analysis set

gCV Geometric coefficient of variation

ICU Intensive care unit

IMP Investigational medicinal product

ITT Intention-to-Treat

LLOQ Lower limit of quantification MAP Mean arterial pressure

Max Maximum

MedDRA Medical dictionary for regulatory activities

Min Minimum

N Number of non-missing values

NLOQ Number of values > lower limit of quantification

PCT Procalcitonine
PK Pharmacokinetic(s)

POD Persistent organ dysfunction

PP Per-protocol
PT Preferred term
Q1 Lower quartile
Q3 Upper quartile
QoL Quality of life

SAP Statistical analysis plan SD Standard deviation

SOFA Score Sequential Organ Failure Assessment Score

t<sub>1/2</sub> Elimination half-lifeV Volume of distribution

|---|---|---|---|
| Statistical Analysis Plan | WI.71.11.0.0. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | 05FEB2020<br>ADR-02 |
| | | | (AdrenOSS-2) |

VAS Visual Analogue Scale

|---------------------------|----------|--------------|
| - W.71.11.0.0. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

## 1. Background and scope

#### As a general rule:

All text copied from the protocol is set in italics type in this statistical analysis plan (SAP).

#### This SAP is based on:

• trial protocol (version 4.1/version 4.2, 07 January 2019/28 August 2019)

#### This SAP covers:

final statistical analysis of the study

The following accompanying documents are part of the SAP:

- Data review plan (AdrenOSS2\_DRP)
- Table shells (AdrenOSS2 Table shells)

An interim analysis was planned and conducted after 28-day follow-up of the first 150 patients was completed. The statistical analysis plan for the interim analysis is not covered in this SAP, but in a separate document.

## 2. Study objectives

#### Primary objective(s):

• To investigate the safety and tolerability of ADRECIZUMAB in patients with early septic shock and elevated bio-ADM (concentration of > 70 pg/ml) in treatment arm A (2 mg/kg) and in treatment arm B (4 mg/kg) over the 90 days study period.

#### Secondary objective(s):

- To obtain first data on efficacy of ADRECIZUMAB in patients with early septic shock and a bio-ADM concentration of > 70 pg/mL in the treatment arms compared with placebo.
- To study the PK of free-ADRECIZUMAB with a focus on plasma accumulation and elimination.

|---------------------------|----------|--------------|
| WI.7 (.1 (. C. C. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

## 3. Study design

## 3.1. Main characteristics of study design

Number of centers: 30 centers in the European Union

Randomized: yes

Blinded: double-blind

Dosing: intravenous infusion (single i.v. dose) over approximately 1 hour

Placebo controlled: yes

Treatments: single i.v. dose of 2 mg/kg Adrecizumab (treatment arm A)

single i.v. dose of 4 mg/kg Adrecizumab (treatment arm B)

single i.v. dose of Placebo (control group)

Randomization ratio: 1:1:2 (treatment arm A : treatment arm B : control group)

PK profile days: Pre-dose

Day 1 (30 min ± 10 min)
Day 2 (24 hours ± 10 hours)
Day 3 (48 hours ± 10 hours)
Day 5 (96 hours ± 10 hours)
Day 7 (144 hours ± 10 hours)
Day 28 (648 hours ± 3 days)

Table 1 Treatment groups and sample sizes

| Treatment | N |
|--------------------------------------|-----|
| Treatment arm A: 2 mg/kg Adrecizumab | 75 |
| Treatment arm B: 4 mg/kg Adrecizumab | 75 |
| Control group: Placebo | 150 |
| Total (randomization ratio 1:1:2) | 300 |

For a flow chart of planned study procedures, please refer to the study protocol.

#### 3.2. Sample Size Determination / Power Analysis

If n=300 early septic shock patients are randomized 1:1 (we assume that both doses can be combined) to placebo and ADRECIZUMAB and assuming that delta SSI is >10%, the power is > 80% to demonstrate an improvement of delta SSI of > 0 with at least 80% probability. The lower bound of the confidence interval will be determined based on the non-parametric Wilcoxon test.

|----------------------|---------------|----------|--------------|
| | WI.71.11.C.O. | Date: | 05FEB2020 |
| Statistical Analysis | Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

The probability of achieving our primary objective, i.e. that the delta SSI is > 0 with at least 80% probability, is 0.87 without interim analysis and 0.85 with the planned interim futility stop.

#### 3.3. Hypotheses

The null-hypothesis is that there is no difference between the Adrecizumab group (both doses combined) and the Placebo group with regard to the primary efficacy endpoint SSI (14 days).

The alternative hypothesis is that the median difference ("delta SSI": Placebo minus Adrecizumab) is larger than zero.

Since confirmative testing is not intended in this phase II trial, a significance level has not been defined.

The study is judged to show a positive result if the lower bound of the two-sided non-parametric 60% confidence interval for delta SSI (Placebo – Adrecizumab) exceeds zero.

## 4. Patient population

The main inclusion criteria are defined as:

- Written informed consent by patient or legally designated representative (according to country-specific regulations)
- Male and female patient, age ≥ 18 years
- Body weight 50 kg 120 kg
- Bio-ADM concentration > 70 pg/ml
- Patient with early septic shock (start of vasopressor therapy < 12 hours)
- Women of childbearing potential must have a negative serum or urine pregnancy test before randomization
- Highly effective method of contraception must be maintained for 6 months after study start by women of childbearing potential and sexually active men
- No care limitation

|----------------------|---------------|----------|--------------|
| | WI.71.11.C.O. | Date: | 05FEB2020 |
| Statistical Analysis | Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## 5. Endpoints for primary and secondary objectives and exploratory endpoints

#### 5.1. Endpoints for primary objectives

#### Safety analysis:

The endpoints for the primary objective are to determine over the 90 days study period:

- Mortality
- Interruption of infusion
- Severity and frequency of treatment-emergent adverse events

#### 5.2. Endpoints for secondary objectives

#### Efficacy analysis:

The primary efficacy endpoint of this study is the

 Sepsis Support Index (SSI) defined as: days with organ support or dead within 14 day follow-up

More precisely: In the time frame of 14 day follow-up, each day on support with vasopressor and/or mechanical ventilation (defined as ventilation received on this day, independent from the duration of mechanical ventilation), and/or renal dysfunction (defined as renal SOFA = 4), or not alive, is counted as 1. The sum over the follow-up period is defined as SSI.

Secondary efficacy endpoints (exploratory) include:

- Sepsis Support Index (SSI) at 28 day follow-up
- Penalized Sepsis Support Index (pSSI) at 14 and 28 day follow-up, defined similar to the SSI with the exception that patients who die get penalized by assigning the maximum value, i.e. the pSSI is set to 14 or 28, respectively
- Persistent organ dysfunction or death at 14 and 28 day follow-up
- Day 28 and day 90 mortality rate
- SSI and pSSI excluding renal component
- SSI weighted for mortality
- Individual Sepsis Support Index components (hemodynamic, respiratory and renal failure) with and without mortality
- Sequential Organ Failure Assessment (SOFA) Score
  - Mean/maximum/total daily SOFA score during stay at ICU
  - Delta SOFA score, defined as maximum versus minimum SOFA during ICU stay
  - Change in SOFA score within 48 hours

|---------------------------|----------|---------------------|
| 141.7 (.1 (.0.0. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | 05FEB2020<br>ADR-02 |
| | | (AdrenOSS-2) |

- SOFA-3 (score limited to cardiovascular, respiratory and renal function)
- Improvement in renal function as change in penKid and creatinine (day 3 day 1, day 7 – day 1)
- Duration of stay at ICU/hospital
- Changes of functional parameters and other parameters during stay at ICU (MAP, creatinine, PaO2/FiO2, blood lactate, MP-pro ADM, inflammatory markers PCT, IL6, DPP3)
- Fluid balance
- Vasopressor use (drug, highest/lowest dose, duration)
- Quality of Life by Euro-QoL-5 (day 28 and day 90)
- Vital signs (heart rate, blood pressure)

## **Endpoints for Pharmacokinetics:**

In sub-study to determine key PK parameters, including:

- peak plasma concentrations (C<sub>max</sub>)
- time to C<sub>max</sub> (t<sub>max</sub>)
- systemic exposure (AUC)
- volume of distribution (V)
- systemic clearance (CL)
- elimination half-life (t<sub>1/2</sub>)

## 5.3. Exploratory endpoints

Not applicable.

#### 6. General conventions

## 6.1. Treatment groups

If not otherwise specified, the following treatment groups will be considered for analysis where applicable and meaningful:

- Adrecizumab 2 mg/kg
- Adrecizumab 4 mg/kg
- Adrecizumab overall (i.e. both Adrecizumab doses)
- Placebo
- Total (i.e. both Adrecizumab doses and Placebo)

|---|---|---|---|
| Statistical Analysis Plan | W.71.11.0.0. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## 6.2. Layout of tables

For numbering of tables, listings and figures, please refer to section 11. Nevertheless, in order to facilitate programming, this numbering might be slightly changed in the final outputs.

Table 2 Layout of tables

| Issue | Specification |
|---|---|
| Basic layout of end-of-text tables and listings (header, footnote) | Titles for all tables, figures, listings: • Study: AdrenOSS-2 (ADR-02) |
| | <ul> <li>Footnotes for all tables, figures, listings include:</li> <li>Program: xxx.sas</li> <li>Generation date: DDMMMYYYY</li> <li>Page X of Y</li> </ul> |
| Font and font size for end-of-text tables and listings | Arial 9 for Tables/Graphs Arial 8 or 9 for Listings Titles in bold and using Arial 10 for Tables and Graphs / Arial 9 or 10 for listings. |
| Text (Title, footnotes, organizational variables and column headers, contents of table) | Case-sensitive, the first letter should be capitalized |
| Subject or Patient as label? | Patient |
| Patient identification numbers | SUBJID (as recorded in eCRF) |
| Categorical Variables | Display of all possible categories (even if a category is not present in the data) In order to increase readability, large tables may also be presented with only the categories observed (e.g. frequency tables for adverse events by primary system organ class, preferred term and severity). |

|---|---|---|---|
| Statistical Analysis Plan | W.71.11.0.0. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

| Issue | Specification |
|---|---|
| In case a category does not occur | Display absolute frequency as "0" |
| Display of percentages in tables: | Aligned by decimal point, one decimal place: • 20.3% • 9.3% • 0.0% • 100.0% |
| Display of units | Presentation case-sensitive and in square brackets, e.g. Concentration [mg/mL] |

#### 6.3. General calculation rules

Data will be listed with the observed number of decimal places. Summary statistics will be presented to the same number of decimal places as the observed data, apart from the means and medians (to one more decimal place), and standard deviations (two more decimal places). Calculated data and summary statistics of calculated data will be presented with an appropriate number of decimal places.

The complete set of summary statistics will be given in case that the number of patients is at least three. For one or two patients, summary statistics will only comprise minimum and maximum.

In case of replicate measurements (e. g. three determinations of a parameter at one planned time-point), means of these measurements will be calculated and will be used for summary statistics without any prior rounding.

Data from unscheduled assessments will only be listed and not presented in summary statistics.

Relative study times and dates will be calculated with respect to the start time and date of the administration of study drug.

|---|---|---|
| WI.71.11.0.0. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | 1.0<br>05FEB2020<br>ADR-02<br>(AdrenOSS-2) |
| | | (AdrenOSS-2) |

Calculation of relative days from onset of adverse events:

The relative day for onset of an adverse event is calculated as "day of onset" minus "day of start of treatment".

#### Duration of adverse events:

The duration of an adverse event (expressed in days) is calculated as "stop date" minus "start date" plus 1.

If parts of the start/stop date of an adverse event are missing (day, month, or year), the relative day for onset and/or the duration of the adverse event are not calculated.

In order to determine if an adverse event or the worsening of an adverse event is a treatment-emergent event, the following rules will be used as a worst case scenario:

- If the date (and time) of onset or change is completely known, the adverse event is considered as treatment-emergent, provided the day (and time) of onset or change is after or on the same day (and time) as first study treatment.
- If the time of onset or change is missing, but the day, month and year is known, the adverse event is considered as treatment-emergent, provided the day of onset or change is after or on the same day as first study treatment, unless other information (e.g. stop date/time) suggest otherwise.
- If the time and day of onset or change is missing, but the month and year is known, the adverse event is considered as treatment-emergent, provided the month of onset or change is after or in the same month as first study treatment, unless other information (e.g. stop date) suggest otherwise.
- If the time, day and month of onset or change is missing, but the year is known, the adverse event is considered as treatment-emergent, provided the year of onset or change is after or in the same year as first study treatment, unless other information (e.g. stop date) suggest otherwise.
- If the time and date of onset or change is completely missing, the adverse event is considered as treatment-emergent, unless other information (e.g. stop date) suggests otherwise.

Calculation of absolute changes from baseline:

• post-dose value - baseline value

Calculation of relative changes from baseline:

• (post-dose value - baseline value)/baseline value

|---|---|---|---|
| Statistical Analysis Plan | W.71.11.0.0. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

Frequencies / percentages for qualitative data:

- Number of observations (frequency)
- Percent

Percentages will be calculated as "frequencies" divided by the number of patients in the population the analysis is based on (i.e. this may include missing data in the denominator).

#### 6.4. Descriptive statistics

Basic descriptive statistics for continuous data comprise:

- Number of observations (N)
- Arithmetic mean
- Standard deviation (SD)
- Minimum (Min)
- Lower quartile (Q1)
- Median
- Upper quartile (Q3)
- Maximum (Max)

<u>Descriptive statistics for continuous variables assumed as log-normally distributed (e. g. PK parameters):</u>

- Number of observations (N)
- Number of observations ≥ LLOQ (NLOQ)
- Arithmetic mean
- Arithmetic SD
- Arithmetic coefficient of variation (CV)
- Geometric mean
- Geometric SD
- Geometric CV(%) (gCV)
- Q1
- Median
- Q3
- Min
- Max

|---------------------------|------|----------|--------------|
| Statistical Analysis Plan | | Date: | 05FEB2020 |
| | Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## 7. Analysis sets and data review criteria

## 7.1. Data sets for analysis

For the determination of patient populations, please refer to the data review plan and the data review protocol. A general definition of data sets for analysis will be:

## Safety analysis set

The safety analysis set includes all patients who

have received study medication.

#### Full analysis set (FAS) (based on intent-to-treat (ITT) principle)

The full analysis set includes all patients who

• have received study medication.

FAS analyses will be done based on the actual treatment ("as treated").

#### Per-protocol (PP) analysis set

The per-protocol analysis set includes all patients who

- are part of the full analysis set
- did receive the study medication according to the protocol with minor deviations only (refer to the Data Review Plan for details)
- satisfy major entry criteria (refer to the Data Review Plan for details).

## Pharmacokinetic analysis set (PKS)

The pharmacokinetic analysis set includes all patients who

- received at least one dose of study medication
- showed sufficient compliance concerning medication, i.e. received the full dose of study medication
- have sufficient concentration PK data to calculate reliable estimates of at least one PK parameter
- are without any protocol violation that would interfere with the interpretation of the PK data.

#### 7.2. Protocol violations/data review

For an overview of checks for identification of protocol violations and data review, please refer to the data review plan.

|---------------------------|------|----------|--------------|
| Statistical Analysis Plan | | Date: | 05FEB2020 |
| | Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## 8. Data analysis

#### 8.1. Statistical software

Statistical analysis will be performed using SAS version 9.3 (or higher) on a Windows 7 (or higher) personal computer. The calculation of pharmacokinetic parameters will be performed with WinNonlin version 8.1.

## 8.2. Definitions, derived variables and handling of missing data

#### 8.2.1. Definitions of time points / time windows

Baseline will be defined per parameter and will be the value/measurement at the following visits:

| Parameter for | Visit |
|-------------------------------|-------------|
| Demographics | Screening 1 |
| Vital signs | Screening 2 |
| ECG | Screening 2 |
| Plasma bio-ADM concentration* | Screening 1 |
| Local laboratory assessment | Screening 2 |
| Arterial blood gas analysis | Screening 2 |
| Biomarker | Day 1 |
| SOFA score | Screening 2 |

<sup>\*</sup> locally measured at study site

#### 8.2.2. Derived variables

#### Extent of exposure:

Extent of exposure will be defined as total exposure in mg and calculated as:

$$total\ exposure\ [mg] = 20\ \frac{mg}{ml}*IMP\ volume\ [ml]*factor$$

where IMP volume is the body weight adjusted IMP volume before addition of NaCl and factor equals 1 for treatment group 4 mg/kg Adrecizumab and ½ for treatment group 2 mg/kg Adrecizumab. Total exposure will not be calculated for the Placebo treatment group.

In case of premature termination of the infusion, total exposure will additionally be multiplied by  $\frac{volume\ administered\ [ml]}{50\ ml}$  in order to account for only partly administration of study drug.



Exposure per kg body weight will be calculated as:

Exposure per 
$$kg$$
 body weight  $\left[\frac{mg}{kg}\right] = \frac{total\ exposure\ [mg]}{body\ weight\ [kg]}$ 

Body mass index (BMI):

$$BMI = \frac{Weight [kg]}{Height [m]^2}$$

#### Sepsis Support Index:

SSI is defined as days with organ support or dead within 14-day follow-up. Organ support days are defined as days with vasopressor, on mechanical ventilation (defined as any mechanical ventilation received on this day, independent from the duration of mechanical ventilation on this day), or need for renal organ support (defined as renal SOFA = 4 (creatinine concentration > 5 mg/dl or > 440  $\mu$ mol/l or urine output < 200ml) due to expected heterogeneity in treatment for renal failure).

The SSI is calculated as follows: In the time frame of 14-day follow-up, each day on support with either vasopressor, and/or mechanical ventilation, and/or need for renal organ support, or not alive, is counted as 1. Patients discharged from the ICU are treated as not receiving any organ support for the days following discharge (unless the patient dies after discharge from ICU: then all days from death to the end of the follow-up period are counted as 1). The sum over the follow-up period is defined as SSI and ranges from 0 to 14.

SSI describes the effect of a given therapy in a pre-defined patient population with septic shock.

SSI calculation will be based on the eCRF entries for Sepsis Support Index (dataset XS). The date of death and the date of discharge from ICU will be derived from the dataset DS (disposition events) and information included for the calculation of the SSI.

## Other versions of the SSI:

- A penalized version of the SSI (pSSI) is defined as above, but including a penalty for patients who die within 14 days: the pSSI is set to 14 for all deaths within 14-day follow-up.
- The individual SSI components will also be compared in the time frame of 14-day follow-up:
  - cardiac component (= sum of days on support with vasopressor)
  - respiratory component (= sum of days with mechanical ventilation)
  - renal failure component (= sum of days with creatinine concentration > 5 mg/dl or > 440 μmol/l or urine output > 200 ml)

|---|---|---|---|
| Statistical Analysis Plan | WI.71.11.0.0. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

death component (= sum of days not alive)

For the cardiac, respiratory and renal failure component patients will only be considered if they survived the respective time period of 14 days.

- A SSI version excluding the renal component will also be evaluated separately in the time frame of 14-day follow-up, so each day on support with either vasopressor, and/or mechanical ventilation, or not alive will be counted as 1.
- A penalized version of the SSI excluding the renal component as defined above.
- A version of the SSI where mortality is given extra weight: Patients being alive during the 14 days' follow up will have an SSI ranging up to 14 (as defined above), while patients who died within that period will be assigned a score of "14 plus the number of days not being alive". Thus the weighted SSI score may range between zero and 28.

The SSI and all other versions of the SSI will also be analyzed for the 28-day follow-up in addition to the 14-day follow-up except for the SSI where mortality is given extra weight (this will only be calculated for the 14-day follow-up).

#### Persistent organ dysfunction (POD) or death:

A novel, composite outcome measure for critical care trials was defined by Heyland et al. (2011):

"We define POD as the persistence of organ dysfunction requiring life-sustaining technologies and it is present when a patient has an ongoing requirement for vasopressors, dialysis, or mechanical ventilation at the outcome assessment points."

Defining renal organ support as renal SOFA = 4 instead of dialysis, the assessed aspects for this endpoint are the same as for the SSI, but at a specific time point instead of within a period.

- Did the patient receive any vasopressor on the outcome assessment day?
- Was patient's creatinine concentration > 5 mg/dl or > 440 μmol/l or was the patient's urine output < 200 ml on the outcome assessment day?
- Did the patient receive mechanical ventilation on the outcome assessment day?
- Was the patient dead at the end of the outcome assessment day (or had the patient already died before)?

The outcome assessment time points will be day 14 and day 28. If one of the questions above is answered with 'Yes' at day 14 or day 28, respectively, the endpoint POD or death will be evaluated as 'Yes' for that patient. If all questions are answered with 'No' or if the patient had already been discharged from ICU, the endpoint will be evaluated as 'No' for that patient, unless the patient died after discharge from ICU.

|---------------------------|----------|--------------|
| | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

#### Sequential Organ Failure Assessment (SOFA) Score:

The SOFA score will be evaluated daily for all patients over the entire stay on ICU (until day 28) or discharge (whatever comes first).

An overview for the determination of the SOFA score can be found Section 13.

For day 1, the last data prior to the treatment has to be used. For this baseline SOFA score only, the renal component will be based on creatinine only (and not on urine output). In the calculation of the score, if multiple values are available within a 24-hour period, the worst value for each parameter will be used, i.e. values resulting in a higher SOFA score will be taken into account. Additionally, parameter values that fall between two scoring intervals will be rounded (e.g. creatinine values to one decimal place) prior to assignment to the categories.

Missing data will not be replaced, i.e. if a single missing value in one of the components occurs, the SOFA score will be set to missing.

Deceased patients will be assigned the maximum SOFA score of 24. In case the patient has been discharged from ICU, the SOFA score will be set to 0 for all days following.

For the cardiovascular system domain, in order to check for vasopressor therapy, the standardized term as allocated during the blinded data review meeting will be used. In case dose information is missing for vasopressor therapy, a dose that would result in the highest SOFA score for the cardiovascular system domain will be assumed.

The change in SOFA score is defined as:

The total SOFA score will be calculated as the sum of daily SOFA scores during the ICU stay for each patient (baseline SOFA will not be considered here).

The mean SOFA score is defined as the total SOFA score divided by the length of stay in the ICU with non-missing SOFA score. The mean score will also be limited to the first 7 days after admission.

The highest SOFA score recorded during the ICU stay will also be recorded. The delta-SOFA score is defined as the difference between the maximum and minimum SOFA score during ICU hospitalization. For these endpoints, the imputed SOFA value for deaths and transferred patients will not be used. Additionally, only non-missing scores will be taken into account in this context. Again, the baseline SOFA will not be considered here.

|---|---|---|---|
| Statistical Analysis Plan | W.71.11.0.0. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

Similar to the full SOFA score, the SOFA-3 score, limited to the cardiovascular, respiratory and renal function, will be calculated including 48 h change, maximum, total, mean and delta (as defined for the full SOFA score).

#### Improvement in renal function:

Improvement in renal function will be determined by analyzing the change in creatinine and penKid at the visits as described below. The following changes will be analyzed for both parameters separately:

- Change from baseline to day 3 (i.e. "Visit 3")
- Change from baseline to day 7 (i.e. "Visit 7")

Missing data due to patient discharge or death will be replaced by carrying the last observation forward, in addition to the analysis using recorded data only.

Measurements will additionally be categorized at baseline and at day 3, respectively, as follows:

| Parameter | Low | High |
|--------------------|-------|-------|
| Creatinine [mg/dL] | ≤ 1.2 | > 1.2 |
| penKid [pmol/L] | ≤ 100 | > 100 |

Patients discharged from ICU or dead will be grouped into the low and high-risk category, respectively.

#### Duration of stay at ICU/hospital:

The duration of stay at ICU will be calculated as:

Duration<sub>(ICU)</sub> = Date of discharge from ICU – Date of ICU admission + 1

The duration of hospital stay will be calculated as:

Duration<sub>(hospital)</sub> = Date of discharge from ICU – Date of hospital admission + 1

In case of missing values, no replacement will be performed.

|---|---|---|---|
| Statistical Analysis Plan | WI.71.11.C.O. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## Changes of functional parameters and other parameters during stay at ICU:

The change from baseline to the last observed (non-missing) value will be analyzed for the following parameters:

- MAP
- PaO<sub>2</sub>/FiO<sub>2</sub>
- Blood lactate
- MR-pro ADM
- PCT
- IL6
- DPP3

The last observed (non-missing) value for fluid balance (calculated as fluid input – fluid output and expressed as absolute value) will be analyzed. In addition, measurements for fluid balance will be categorized as follows:

| Parameter | Low | High |
|------------------------|--------|--------|
| Fluid balance [ml/day] | ≤ 1000 | > 1000 |

#### Vasopressor use:

Vasopressor use will be analyzed as frequency tables by drug (ATC code) and number of vasopressors used, highest and lowest dose (per ATC code) as well as mean duration of vasopressor use expressed as days and summarized by treatment group and ATC code using descriptive summary statistics. In case of ongoing vasopressor use, the end date will be replaced by the date of discharge from ICU or the date of death (whatever occurs first). In case dose information of vasopressor use is given in different units, it will be converted to one common unit. The conversion factors are discussed during the blinded data review meeting.

#### Quality of Life by Euro-QoL-5:

Quality of Life will be measured by Euro-QoL-5 questionnaire and analyzed for discharge from ICU, follow-up day 28 and follow-up day 90, respectively.

In addition to the possible answers (i.e. level 1-5), the single dimensions will be dichotomized into 'no problems' (i.e. level 1) and 'problems' (i.e. level 2-5).

|------------|---------------------------|----------|--------------|
| WI.A.IX.O. | WI.7 1.11.0.0. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

Change in quality of life expressed by visual analogue scale (VAS) will be defined as:

- VAS at discharge from ICU VAS at day 90
- VAS at day 28 VAS at day 90.

The VAS will be analyzed by treatment group and visit in addition to the changes as defined above.

## Vital signs:

The change in vital signs (heart rate, systolic and diastolic blood pressure as well as MAP) will be analyzed for the visits as described below. The following changes will be analyzed for the mentioned parameters separately:

- Change from baseline to day 3
- Change from baseline to day 7

Missing data due to patient discharge or death will be replaced by carrying the last observation forward, in addition to the analysis using reported data only.

Measurements will additionally be categorized at baseline and at day 3, respectively, for MAP and heart rate as follows:

| Parameter | Low | High |
|------------------|-------|-------|
| MAP [mmHg] | ≤ 65 | > 65 |
| Heart rate [bpm] | ≤ 100 | > 100 |

Missing values for patients discharged from ICU or dead will be grouped into the low and high-risk category, respectively.

#### **APACHE II score**

For an overview of the single items for the derivation of the APACHE II score, please see Section 13.

The item 'Temperature' should be measured rectal according to the scoring table, but is only available as oral/tympanic in this study. Nevertheless, it will be used without applying a correction factor for this item.



The parameter A-a Gradient is needed to score the item 'Oxygenation'. As it was not recorded in this study, it will be derived as:

A-a  $_{O2}$  Gradient = [ (FiO<sub>2</sub>) × (Atmospheric Pressure - H<sub>2</sub>O Pressure) - (PaCO<sub>2</sub>/0.8) ] – PaO<sub>2</sub>

The following reference values will be used to calculate the A-a  $_{\rm O2}$  Gradient:

Atmospheric pressure: 760 mmHg

H<sub>2</sub>O pressure: 47 mmHg

PaCO<sub>2</sub>: 40 mmHg

In case the calculation for the A-a  $_{\rm O2}$  Gradient results in a negative value, it will be set to 0. The single item score for 'Serum creatinine' needs to be doubled for acute renal failure. In this context, all patients with 'Chronic Renal Disease' or 'Hemodialysis' marked 'Yes' on the medical history (non cardiovascular co-morbidities) page in the eCRF will be defined as no acute renal failure patients (i.e. the score will be doubled for all other patients).

For all parameters used to derive the APACHE II score, the value measured/determined at Screening will be used. Only in case this value is missing, the value of Day 1 will be taken into account irrespective of if it was measured/determined before or after IMP administration (as this sometimes is not obvious from the data recorded). This is justified by medical experience stating that values do not vary significantly within such a short time frame (around 24 hours).

Values that fall between two single item scores will be rounded to the number of decimals specified for the respective item and classified accordingly.

The APACHE II score ranges from 0 to 71.

## PaO<sub>2</sub>/FiO<sub>2</sub> ratio

The PaO<sub>2</sub>/FiO<sub>2</sub> ratio as recorded in the eCRF will not be used in any analyses due to unclear unit information. It will be recalculated based on the recorded values for PaO<sub>2</sub> and FiO<sub>2</sub> as follows:

$$\frac{PaO_2}{FiO_2}[mmHg] = \frac{PaO_2[mmHg]}{\left(\frac{FiO_2[\%]}{100}\right)}$$

This applies to all visits where only a single value is recorded. No recalculation will be performed for visits where minimum and maximum values had to be documented. The (recalculated) value for the ratio will be set to missing in this case.

|---------------------------|----------|--------------|
| Statistical Analysis Plan | Date: | 05FEB2020 |
| | Project: | ADR-02 |
| | | (AdrenOSS-2) |

In case  $FiO_2$  < 1 was recorded, this value will be multiplied by 100 to achieve % values, irrespectively of the unit provided by the sites.

PaO<sub>2</sub> values recorded in kPa will be multiplied by 7.5 in order to obtain values in mmHg.

#### 8.2.3. Handling of missing values

If not already specified in section 8.2.2 for the single endpoints, the following rules for handling of missing values will be applied:

If the SSI is already well-defined despite missing data, i.e. the SSI contribution for a specific day is 1 despite a missing component (e.g. creatinine is missing, but patient received mechanical ventilation), it will not be treated as missing. However, all missing data within each component will be discussed during the blinded data review.

Other replacement of missing values will not be performed.

Data from patients who prematurely terminate the trial will be used to the maximum possible extent.

#### 8.3. Sensitivity analyses

Sensitivity analyses will be performed for the following sub-populations of FAS:

- a) exclusion of the first 2 patients from every center (according to the date of dosing)
- b) inclusion of centers who had randomized at least 4 patients
- c) inclusion of patients with a DPP3 concentration ≤ 70 ng/mL at baseline.

The following endpoints will be analyzed for these subgroups: SSI (follow-up until Day 14), mortality at Day 28 and Day 90 using FAS.

#### 8.4. Disposition

An overview of all patients who entered the study, who were randomized and who completed the study will be provided by treatment group and overall. Reasons for all post-randomized discontinuations will be given by treatment group.

Furthermore, an overview of all patients who are in the different analysis sets will be provided by treatment group.

|---------------------------|----------|--------------|
| <br>WI.7 (.1 (. O. O. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | _ | (AdrenOSS-2) |

#### 8.5. Demographic data and baseline characteristics

Demographic data and baseline characteristics will be summarized for the safety analysis set.

#### Demographic data and baseline characteristics

Summary statistics will be presented for age, weight, height, BMI, vital signs at screening (body temperature, heart rate, MAP, systolic and diastolic blood pressure, respiratory rate), creatinine, blood lactate, SOFA score, APACHE II score, bio-ADM concentration. Frequency tables for qualitative data (gender, ethnic origin, origin of sepsis, location before ICU admission) will be provided.

In order to check structural comparison of the three treatment groups, the Kruskal-Wallis test will be performed for continuous baseline characteristics.

Categorical variables will be compared using the Chi<sup>2</sup> test for contingency tables.

#### Medical history

Frequency tables of medical history data by treatment group will be provided using MedDRA coding (Version 22.1) and differentiating between past and ongoing diseases as well as between cardiovascular and non-cardiovascular co-morbidities and other medical history present at inclusion.

#### Prior and concomitant medications

Frequency tables for prior and/or concomitant medications will be presented by treatment group taking WHO classification into account. Prior medications are medications which started and ended prior to study drug administration. Concomitant medications are defined as all recorded medications not classified as prior medication.

## Physical examination

Results of the physical examination (normal, clinically significant, clinically not significant) will be presented as frequency tables by treatment groups.

#### Diagnosis of early septic shock

MAP [mmHg] before and after fluid resuscitation, volume administered [ml] for fluid resuscitation and plasma bio-ADM concentration [pg/ml] will be analyzed in the context of diagnosis of early septic shock by descriptive summary statistics.

Refractoriness to fluid resuscitation (yes, no) will be presented using frequency tables.

|----------------------|---------------------------|----------|--------------|
| | Statistical Analysis Plan | Date: | 05FEB2020 |
| Statistical Analysis | | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## 8.6. Analysis of primary endpoints

The analyses of the endpoints for safety and tolerability will be performed on the safety analysis set.

All efficacy analyses will be performed on the full analysis set. In addition, analyses will be presented for the per-protocol set.

#### Severity and frequency of treatment-emergent adverse events:

The absolute number of treatment-emergent adverse events as well as the number of patients with treatment-emergent adverse events will be analyzed using frequency tables by treatment group. An analysis by Primary System Organ Class (SOC) and Preferred Term (PT) will be given as well. These frequencies will be given for all treatment-emergent adverse events as well as by severity grade (mild (grade 1), moderate (grade 2), severe (grades  $\geq$  3)).

95% confidence intervals will be calculated for adverse event incidences by treatment group applying the Clopper-Pearson method for each SOC and each PT.

#### Mortality:

All-cause mortality for 90-day follow-up will be evaluated using Kaplan-Meier plots comparing Adrecizumab (doses combined) vs. Placebo, and Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg vs. Placebo (each with log-rank test without adjustment).

In addition, frequency tables will be provided for all-cause mortality by treatment group. Separate tables will be provided for all-cause mortality during 28-day and 90-day follow-up.

#### <u>Interruption of infusion:</u>

The number of patients with at least one interruption of infusion as well as the number of interruptions will be analyzed using frequency tables. In case the infusion was stopped prematurely, this will be given as a separate category in the frequency tables.

The three treatment groups will be compared by the Chi<sup>2</sup> statistic with regard to the categories "complete infusion" and "infusion interrupted at least once or stopped prematurely".

## Sepsis Support Index (SSI) within 14 days:

The primary analysis for efficacy will be based on combining both Adrecizumab doses and comparing the treated groups versus the Placebo group and performed on the FAS. A second-line analysis will compare the two doses separately versus Placebo for differences in efficacy.

|---------------------------|----------|--------------|
| W.7 (.1 (. O. O. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

For the primary efficacy endpoint, a non-parametric 60% confidence interval will be calculated for the difference between Adrecizumab (doses combined) and Placebo using the Hodges-Lehmann estimator. Testing for differences between treatment groups will be performed by applying the Kolmogorov-Smirnov test. The empirical cumulative distribution functions will be graphically displayed.

The analysis described above will also be applied for comparing Adrecizumab 2 mg/kg vs. Placebo, and Adrecizumab 4 mg/kg vs. Placebo.

Summary statistics of the SSI by treatment group and histograms for each group will also be prepared.

## 8.7. Analysis of secondary endpoints

All efficacy analyses will be performed on the full analysis set. In addition, analyses will be presented for the per-protocol set.

#### Mortality:

All-cause mortality 28-day follow-up will be evaluated using Kaplan-Meier plots comparing Adrecizumab vs. Placebo and Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg vs. Placebo (each with log-rank test without adjustment).

An additional analysis will include Cox regression modelling concerning 28-days as well as 90-days mortality, uni- and multivariate, including covariates to adjust for potential confounders. Potential confounders comprise baseline characteristics with a p-value < 0.1 determined during the analyses for structural comparison of baseline characteristics.

If not otherwise specified, baseline values of the above mentioned covariates will be used and it will be assumed that covariates do not vary during follow-up time.

In this context, the following models with only one covariate will be fitted (SAS syntax):

```
PROC PHREG DATA=[...];

CLASS treatment cat_var;

MODEL days*survive(0) = treatment <cat_var or cont_var>;

RUN;
```

where days is the survival time in days, survive is the censoring variable with 0 indicating censoring, treatment is the treatment group (1= Adrecizumab, 0=Placebo), cat\_var or cont var is the respective categorical or continuous covariate.

|----------------------|---------------------------|----------|--------------|
| | Statistical Analysis Plan | Date: | 05FEB2020 |
| Statistical Analysis | | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

The proportional hazards assumption will be checked graphically by plotting log(-log(S(t))) vs. t, i.e. by looking for parallelism with regard to treatment group and categorical covariates. The survival curve S(t) is estimated by the Kaplan-Meier method.

Multivariate modelling will include all covariates mentioned above as well as treatment:

```
PROC PHREG DATA=[...];

CLASS treatment cat_vars;

MODEL days*survive(0) = treatment all_vars;

RUN;
```

with treatment (1= Adrecizumab, 0=Placebo) and with all\_vars representing all categorical and continuous variables mentioned above.

#### Other versions of the SSI:

The other versions of the SSI will be analyzed using the same methods and procedures as described for the primary efficacy endpoint.

#### Persistent organ dysfunction or death at 14- and 28-day follow-up:

This dichotomous endpoint will be analyzed via cross-tables (2 by 2) for Adrecizumab vs. Placebo including Chi² test. In addition, 2 by 3 tables for Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg vs. Placebo will be presented together with the results of a Cochran-Armitage test for trend.

#### SOFA score:

Descriptive summary statistics will be presented for the SOFA score and SOFA-3 score by time point as well as for the defined endpoints: SOFA<sub>change</sub>, total score, mean score (over entire ICU stay), mean score (over first 7 days of ICU stay), maximum SOFA score during ICU stay, delta-SOFA score (the difference between the maximum and minimum SOFA score during ICU stay).

The Kruskal-Wallis test will be applied for the defined endpoints to compare Adrecizumab 2mg/kg vs. Adrecizumab 4 mg/kg vs. Placebo. Pairwise comparison (each Adrecizumab dose vs. Placebo) will be carried out using the Wilcoxon test.

|---------------------------|----------|--------------|
| | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

#### Improvement in renal function:

Improvement in renal function will be analyzed using descriptive summary statistics. Analyses for absolute values as well as the changes as defined above will be presented in this context.

The following endpoints are considered:

Change in penKid (day 3 – day 1), change in penKid (day 7 – day 1), Change in creatinine (day 3 – day 1), change in creatinine (day 7 – day 1)

The Kruskal-Wallis test will be applied for these endpoints to compare Adrecizumab 2mg/kg vs. Adrecizumab 4 mg/kg vs. Placebo. Pairwise comparison (each Adrecizumab dose vs. Placebo as well as Adrecizumab (combined doses) vs. Placebo) will be carried out using the Wilcoxon test.

#### **Duration of stay in ICU/hospital:**

The duration of stay in ICU as well as the duration of stay in hospital will be analyzed using descriptive summary statistics.

The Kruskal-Wallis test will be applied to compare Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg vs. Placebo. Pairwise comparison (each Adrecizumab dose vs. Placebo) will be carried out using the Wilcoxon test.

## Changes of functional parameters and other parameters during stay at ICU:

MAP (minimum, maximum), creatinine, PaO2/FiO2 (minimum, maximum), blood lactate, fluid balance, bio-ADM, MR-proADM, PCT, IL6, penKid, DPP3, vr-hGH) will be evaluated using descriptive summary statistics by treatment group and time point (Day 1, Day 2, Day 3 etc.).

#### Vasopressor use:

Continuous variables for vasopressor use will be analyzed by descriptive summary statistics; categorical variables analyses will be carried out using frequency tables.

#### Quality of Life by Euro-Qol-5:

The VAS for Euro-Qol-5 will be analyzed by descriptive summary statistics. The change from discharge from ICU and from follow-up day 28 to the assessment at 90-day follow-up will also be analyzed by descriptive summary statistics.

|---------------------------|----------|--------------|
| Statistical Analysis Plan | Date: | 05FEB2020 |
| | Project: | ADR-02 |
| | | (AdrenOSS-2) |

The single dimensions of the questionnaire (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) will be presented using frequency tables for all possible answers.

#### Vital signs:

Vital signs as described in section 8.2.2 will be analyzed using descriptive summary statistics and frequency tables.

#### 8.8. Pharmacokinetic data analyses

PK samples from 80 patients will be collected at designated sites participating in the PK substudy.

The analyses of Adrecizumab plasma concentrations and derived PK parameters will be performed on the PKS.

The PK parameters will be analyzed by descriptive summary statistics.

#### 8.8.1. Pharmacokinetic parameters

The following parameters will be determined from the individual plasma concentration-time profiles of Adrecizumab using noncompartmental methods based on actual relative sampling times:

#### **Definitions of pharmacokinetic parameters**

| AUC <sub>0-last</sub> | Systemic exposure | e. i.e. area ur | nder the observed | concentration-time curve |
|---|---|---|---|---|

from time zero up to the last time point with quantifiable plasma

concentration (t<sub>last</sub>). The area will be calculated according to the linear

up/log down trapezoidal rule.

AUC<sub>0-144h</sub> Area under the observed concentration-time curve from time zero up to

144 h. The area will be calculated according to the linear up/log down

trapezoidal rule.

C<sub>max</sub> Observed maximum concentration

 $t_{max}$  Observed time of maximum concentration  $C_{max}$ 

C<sub>last</sub> Last observed concentration

 $t_{\text{last}} \hspace{1.5cm} \text{Time of last observed concentration } C_{\text{last}}$ 

t<sub>1/2</sub> Terminal elimination half-life
|---------------------------|----------|--------------|
| Statistical Analysis Plan | Date: | 05FEB2020 |
| | Project: | ADR-02 |
| | | (AdrenOSS-2) |

CL Systemic clearance
V Volume of distribution

Single concentration data will be shown with the significant number of decimal places as provided by the analytical lab. Derived parameters, as far as they do not present single concentrations such as  $C_{\text{max}}$ , will be listed with an appropriate number of significant digits (at least 3).

Exposure parameters ( $C_{max}$  and  $AUC_{0-last}$ ) will also be dose-normalized (i.e. divided by dose) for the investigation of dose-dependency.

## 8.8.2. Analysis of pharmacokinetic endpoints

Not applicable.

## 8.8.3. Descriptive pharmacokinetic analyses

The PK analysis will be performed for both active treatment groups.

The individual time courses of the plasma concentrations of Adrecizumab will be listed and summarized descriptively by treatment group and time point.

Summary statistics by time point will be calculated including only those samples which were taken according to the pre-defined sampling schedule, i.e.: 30 min  $\pm$  10 min, 24 h  $\pm$  10 h, 48 h  $\pm$  10 h, 96 h  $\pm$  10 h, 144 h  $\pm$  10 h, 28 d  $\pm$  3 d.

For the calculation of summary statistics a data point below the lower limit of quantification (LLOQ) will be substituted by an estimated value of half the lower limit of quantification (½ LLOQ). However, means, standard deviations and coefficients of variation at any time-point will only be calculated if at least 2/3 of the individual data had been measured and were above the lower limit of quantification. In tables showing mean values, where values below LLOQ are included in the calculation of mean values, these means will be marked.

Individual plasma concentration-time profiles will be plotted for Adrecizumab (up to 8 profiles in one plot) for each dose group considering all patients with available PK concentration data even if not included in the PKS using actual relative sampling times. Geometric means of Adrecizumab plasma concentrations including one SD range will be plotted for both active treatment groups in one plot (for PKS). Individual and geometric mean concentration versus time curves will be plotted using both linear and semi-logarithmic scaling.

|---------------------------|----------|--------------|
| Statistical Analysis Plan | Date: | 05FEB2020 |
| | Project: | ADR-02 |
| | | (AdrenOSS-2) |

Summary statistics will be calculated for each pharmacokinetic parameter by dose group based on PKS.

# 8.9. Pharmacodynamic data analyses

There are no study variables specifically classified as pharmacodynamics endpoints.

## 8.10. Evaluation of relationships between endpoints

The Cox regression model will be applied to investigate the effects of potential confounders on 90-days mortality. Details are described in Section 8.7.

# 8.11. Safety analysis

All safety analyses described below will be based on the Safety Analysis Set and will only be exploratory.

### 8.11.1. Extent of exposure

Total exposure [mg] and relative exposure [mg/kg] will be analyzed by descriptive summary statistics.

#### 8.11.2. Adverse events

An overview over all adverse events (original term as well as SOC and PT) will be generated as patient data listings, including onset relative to start of treatment, duration, intensity, seriousness and relationship to the study drug, action taken and outcome.

The incidence of treatment-emergent adverse events as well as number of patients with treatment-emergent adverse events will be summarized by SOC, PT and relationship to the study drug (certain, probable/likely, possible, unlikely, unrelated) for all treatment groups.

Treatment emergent events are adverse events not present at baseline, or adverse events that worsened after start of treatment even if they were present at baseline.

Deaths and serious adverse events will be listed separately (if applicable).

|----------------------|---------------------------|----------|--------------|
| | Statistical Analysis Plan | Date: | 05FEB2020 |
| Statistical Analysis | | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

## 8.11.3. Clinical laboratory

Complete listings for laboratory values (hematology, biochemistry) will be generated. Laboratory values outside the normal range will be marked.

Only values  $\geq 0$  will be included in statistical evaluations.

Results from laboratory tests will be summarized by treatment group and time point using descriptive summary statistics including changes from baseline. Since different local labs were involved in this trial with different normal ranges, the laboratory results will be standardized to the normal range prior to analysis, i.e. a value X will be transformed to:

Y = (X - LLN) / (ULN - LLN), where LLN and ULN denote lower limit of normal and upper limit of normal, respectively.

Extreme relative changes (for original laboratory values) from baseline to follow-up visits (post minus baseline) will be categorized as:

Maximum increase from baseline: (maximum value post – baseline) / baseline

 $\geq 1.5, \geq 2.0$ 

Maximum decrease from baseline: (baseline - minimum value post) / baseline  $\geq 0.5$ 

A frequency table by treatment will be generated for these categorized changes.

In addition, changes from "from within normal range to above normal range" will be evaluated and categorized as:

"changes to at least 1.5-time upper limit normal", "changes to at least twice upper limit normal".

A frequency table by treatment will be generated for these categorized changes from normal at baseline.

## 8.11.4. Vital signs and body temperature

Minimum and maximum values for vital signs assessed within one day will be analyzed using descriptive summary statistics (including changes from baseline) by treatment group and time point (Day 1, Day 2, Day 3 etc.), i.e. concerning body temperature, heart rate, systolic and diastolic blood pressure as well as respiratory rate and MAP.

Only values > 0 will be included in summary statistics.

### 8.11.5. ECG

Frequencies of overall interpretation (normal, abnormal and clinically not significant, abnormal and clinically significant) will be tabulated by treatment group and time point.

|----------------------|---------------------------|----------|--------------|
| | Statistical Analysis Plan | Date: | 05FEB2020 |
| Statistical Analysis | | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

#### 8.11.6. Biomarker

Biomarker results will be analyzed by descriptive summary statistics for the different scheduled determination time points as well as expressed as changes from baseline.

#### 8.11.7. Other assessments

For all other safety data (e.g. echocardiography) listings will be generated.

Patient data listings will also be provided in case derived variables are used for analysis (e.g. for SSI score, SOC and PT for medical history terms or duration of adverse events). A detailed overview of listings to be provided in this context can be found in section 11.

# 9. Changes to the protocol

"SSI weighted for mortality" has been defined as additional secondary endpoint.

In addition, the Kolmogorov-Smirnov test will be performed for the primary efficacy endpoint.

# 10. Changes to the SAP after finalization

Not applicable.

|---------------------------|----------|--------------|
| WI.71.11.C.O. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

# 11. Contents of statistical tables and figures

| | | | 14 Tables and figures referred to but not included in the |
|---|---|---|---|
| | | | text |
| | | | 14.1 Demographic data and general study information |
| * | Table | 14.1-1 | Overview of patients |
| | Table | 14.1-2 | Reasons for post-randomized discontinuations |
| * | Table | 14.1-3 | Patients in the different analysis sets |
| | Listing | 14.1-4 | Patients in the different analysis sets |
| * | Table | 14.1-5 | Demographic data (descriptive summary statistics) |
| | Table | 14.1-6 | Structural comparison of baseline characteristics (continuous variables) |
| * | Table | 14.1-7 | Demographic data (frequency tables) |
| | Table | 14.1-8 | Structural comparison of baseline characteristics (categorical variables) |
| | Table | 14.1-9 | Medical history (frequency tables) |
| | Listing | 14.1.10 | Overview of medical history |
| | Table | 14.1-11 | Prior and concomitant medications (frequency tables) |
| | Listing | 14.1.12 | Overview of prior and concomitant medications |
| | Table | 14.1-13 | Physical examination (frequency tables) |
| | Table | 14.1-14 | Diagnosis of early septic shock (descriptive summary statistics) |
| | Table | 14.1-15 | Diagnosis of early septic shock (frequency tables) |
| | | | 14.2 Analysis of primary and secondary endpoints |
| | | | 14.2.1 Analysis of primary endpoints |
| | | | 14.2.1.1 Mortality |
| * | Figure | 14.2.1.1-1 | Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab) |
| | Figure<br>Figure | 14.2.1.1-1<br>14.2.1.1-2 | 1 |
| | | | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group |
| * | | | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| * | Figure | 14.2.1.1-2 | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) 14.2.1.2 Interruption of infusion |
| * | Figure<br>Table | 14.2.1.1-2 | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) 14.2.1.2 Interruption of infusion Frequencies for interruption of infusion |
| * | Figure<br>Table | 14.2.1.1-2 | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) 14.2.1.2 Interruption of infusion Frequencies for interruption of infusion Comparison of treatment groups for interruption of infusion 14.2.1.3 Severity and frequency of treatment-emergent |
| * | Figure Table Table | 14.2.1.1-2<br>14.2.1.2-1<br>14.2.1.2-2 | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) 14.2.1.2 Interruption of infusion Frequencies for interruption of infusion Comparison of treatment groups for interruption of infusion 14.2.1.3 Severity and frequency of treatment-emergent adverse events Frequencies for treatment-emergent adverse events by SOC, |
| * | Figure Table Table Table | 14.2.1.1-2<br>14.2.1.2-1<br>14.2.1.2-2<br>14.2.1.3-1 | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) 14.2.1.2 Interruption of infusion Frequencies for interruption of infusion Comparison of treatment groups for interruption of infusion 14.2.1.3 Severity and frequency of treatment-emergent adverse events Frequencies for treatment-emergent adverse events by SOC, PT and severity Clopper-Pearson confidence interval for treatment-emergent adverse events 14.2.1.4 Sepsis Support Index (SSI) within 14 days |
| * | Figure Table Table Table | 14.2.1.1-2<br>14.2.1.2-1<br>14.2.1.2-2<br>14.2.1.3-1 | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) 14.2.1.2 Interruption of infusion Frequencies for interruption of infusion Comparison of treatment groups for interruption of infusion 14.2.1.3 Severity and frequency of treatment-emergent adverse events Frequencies for treatment-emergent adverse events by SOC, PT and severity Clopper-Pearson confidence interval for treatment-emergent adverse events 14.2.1.4 Sepsis Support Index (SSI) within 14 days Sepsis Support Index (incl. different variations of SSI) |
| * | Figure Table Table Table Table | 14.2.1.1-2<br>14.2.1.2-1<br>14.2.1.2-2<br>14.2.1.3-1<br>14.2.1.3-2 | (Placebo vs. Adrecizumab) Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) 14.2.1.2 Interruption of infusion Frequencies for interruption of infusion Comparison of treatment groups for interruption of infusion 14.2.1.3 Severity and frequency of treatment-emergent adverse events Frequencies for treatment-emergent adverse events by SOC, PT and severity Clopper-Pearson confidence interval for treatment-emergent adverse events 14.2.1.4 Sepsis Support Index (SSI) within 14 days |

|--------|---------------------------|----------|--------------|
| $\neg$ | WI.A.IV.O.O. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

| * | Figure | 14.2.1.4-4 | Histogram for SSI within 14 days (Placebo vs. Adrecizumab) |
|---|---|---|---|
| * | Figure | 14.2.1.4-5 | Histogram for SSI within 14 days (Placebo vs. Adrecizumab 2 |
| | | | mg/kg vs. Adrecizumab 4 mg/kg) |
| | | | 14.2.2 Analysis of secondary endpoints |
| | | | 14.2.2.1 Mortality |
| * | Figure | 14.2.2.1-1 | Kaplan-Meier plot for 28-day follow-up by treatment group (Placebo vs. Adrecizumab) |
| * | Figure | 14.2.2.1-2 | Kaplan-Meier plot for 28-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| | Table | 14.2.2.1-3 | Cox regression |
| | | | 14.2.2.2 Other versions of the SSI |
| | Table | 14.2.2.2-1 | Descriptive summary statistics for SSI within 28 days |
| | Figure | 14.2.2.2-2 | Histogram for SSI within 28 days (Placebo vs. Adrecizumab) |
| | Figure | 14.2.2.2-3 | Histogram for SSI within 28 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| * | Table | 14.2.2.2-4 | Descriptive summary statistics for pSSI within 14 days |
| * | Figure | 14.2.2.2-5 | Histogram for pSSI within 14 days (Placebo vs. Adrecizumab) |
| * | Figure | 14.2.2.2-6 | Histogram for pSSI within 14 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| | Table | 14.2.2.2-7 | Descriptive summary statistics for pSSI within 28 days |
| | Figure | 14.2.2.2-8 | Histogram for pSSI within 28 days (Placebo vs. Adrecizumab) |
| | Figure | 14.2.2.2-9 | Histogram for pSSI within 28 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| * | Table | 14.2.2.2-10 | Descriptive summary statistics for SSI cardiac component within 14 days |
| * | Figure | 14.2.2.2-11 | Histogram for SSI cardiac component within 14 days (Placebo vs. Adrecizumab) |
| * | Figure | 14.2.2.2-12 | Histogram for SSI cardiac component within 14 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| | Table | 14.2.2.2-13 | Descriptive summary statistics for SSI cardiac component within 28 days |
| | Figure | 14.2.2.2-14 | Histogram for SSI cardiac component within 28 days (Placebo vs. Adrecizumab) |
| | Figure | 14.2.2.2-15 | Histogram for SSI cardiac component within 28 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| * | Table | 14.2.2.2-16 | Descriptive summary statistics for SSI respiratory component within 14 days |
| * | Figure | 14.2.2.2-17 | Histogram for SSI respiratory component within 14 days (Placebo vs. Adrecizumab) |
| * | Figure | 14.2.2.2-18 | Histogram for SSI respiratory component within 14 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| | Table | 14.2.2.2-19 | Descriptive summary statistics for SSI respiratory component within 28 days |
| | Figure | 14.2.2.2-20 | Histogram for SSI respiratory component within 28 days (Placebo vs. Adrecizumab) |

|--------|---------------------------|----------|--------------|
| $\neg$ | WI.A.IV.O.O. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

| Т | | |
|---|---|---|
| Figure | 14.2.2.2-21 | Histogram for SSI respiratory component within 28 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Table | 14.2.2.2-22 | Descriptive summary statistics for SSI renal failure component within 14 days |
| · · | 14.2.2.2-23 | Histogram for SSI renal failure component within 14 days (Placebo vs. Adrecizumab) |
| Figure | 14.2.2.2-24 | Histogram for SSI renal failure component within 14 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Table | 14.2.2.2-25 | Descriptive summary statistics for SSI renal failure component within 28 days |
| Figure | 14.2.2.2-26 | Histogram for SSI renal failure component within 28 days (Placebo vs. Adrecizumab) |
| Figure | 14.2.2.2-27 | Histogram for SSI renal failure component within 28 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Table | 14.2.2.2-28 | Descriptive summary statistics for SSI death component within 14 days |
| Figure | 14.2.2.2-29 | Histogram for SSI death component within 14 days (Placebo vs. Adrecizumab) |
| Figure | 14.2.2.2-30 | Histogram for SSI death component within 14 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Table | 14.2.2.2-31 | Descriptive summary statistics for SSI death component within 28 days |
| Figure | 14.2.2.2-32 | Histogram for SSI death component within 28 days (Placebo vs. Adrecizumab) |
| Figure | 14.2.2.2-33 | Histogram for SSI death component within 28 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Table | 14.2.2.2-34 | Descriptive summary statistics for SSI within 14 days excl. renal component |
| Figure | 14.2.2.2-35 | Histogram for SSI within 14 days excl. renal component (Placebo vs. Adrecizumab) |
| Figure | 14.2.2.2-36 | Histogram for SSI within 14 days excl. renal component (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Table | 14.2.2.2-37 | Descriptive summary statistics for SSI within 28 days excl. renal component |
| Figure | 14.2.2.2-38 | Histogram for SSI within 28 days excl. renal component (Placebo vs. Adrecizumab) |
| Figure | 14.2.2.2-39 | Histogram for SSI within 28 days excl. renal component (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Table | 14.2.2.2-40 | Descriptive summary statistics for pSSI within 14 days excl. renal component |
| Figure | 14.2.2.2-41 | Histogram for pSSI within 14 days excl. renal component (Placebo vs. Adrecizumab) |
| Figure | 14.2.2.2-42 | Histogram for pSSI within 14 days excl. renal component (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Table | 14.2.2.2-43 | Descriptive summary statistics for pSSI within 28 days excl. renal component |
| | Figure Figure Table Figure Table Figure Table Figure Table Figure Table Figure Table Figure Table Figure Figure Table Figure Figure Figure Figure Figure | Table 14.2.2.2-22 Figure 14.2.2.2-24 Figure 14.2.2.2-25 Table 14.2.2.2-26 Figure 14.2.2.2-27 Table 14.2.2.2-27 Table 14.2.2.2-28 Figure 14.2.2.2-30 Table 14.2.2.2-31 Figure 14.2.2.2-31 Figure 14.2.2.2-32 Figure 14.2.2.2-34 Figure 14.2.2.2-35 Figure 14.2.2.2-36 Table 14.2.2.2-37 Figure 14.2.2.2-38 Figure 14.2.2.2-39 Table 14.2.2.2-40 Figure 14.2.2.2-41 Figure 14.2.2.2-42 |

|--------|---------------------------|----------|--------------|
| $\neg$ | WI.A.N.O.O. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

| | Figure | 14.2.2.2-44 | Histogram for pSSI within 28 days excl. renal component (Placebo vs. Adrecizumab) |
|---|---|---|---|
| | Figure | 14.2.2.2-45 | Histogram for pSSI within 28 days excl. renal component (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| | Table | 14.2.2.2-46 | Descriptive summary statistics for SSI within 14 days where mortality is given extra weight |
| * | Figure | 14.2.2.2-47 | Histogram for SSI within 14 days where mortality is given extra weight (Placebo vs. Adrecizumab) |
| * | Figure | 14.2.2.2-48 | Histogram for SSI within 14 days where mortality is given extra weight (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| | | | 14.2.2.3 Persistent organ dysfunction or death at 14- and 28-day follow-up |
| | Table | 14.2.2.3-1 | Persistent organ dysfunction or death (Placebo vs. Adrecizumab) |
| | Table | 14.2.2.3-2 | Persistent organ dysfunction or death (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| | | | 14.2.2.4 SOFA score |
| | Table | 14.2.2.4-1 | Descriptive summary statistics for SOFA score |
| | Table | 14.2.2.4-2 | Descriptive summary statistics for SOFA-3 score |
| | | | 14.2.2.5 Improvement in renal function |
| | Table | 14.2.2.5-1 | Descriptive summary statistics for improvement in renal function |
| | Table | 14.2.2.5-2 | Frequency tables for improvement in renal function |
| | | | 14.2.2.6 Duration of stay in ICU/hospital |
| | Table | 14.2.2.6-1 | Descriptive summary statistics for stay in ICU/hospital |
| | | | 14.2.2.7 Changes of functional parameters and other parameters during stay at ICU |
| | Table | 14.2.2.7-1 | Descriptive summary statistics for functional and other parameters during stay at ICU |
| | Table | 14.2.2.7-2 | Frequencies tables for fluid balance |
| | | | 14.2.2.8 Vasopressor use |
| | Table | 14.2.2.8-1 | Frequency tables for vasopressor use |
| | Table | 14.2.2.8-2 | Descriptive summary statistics for vasopressor use |
| | | | 14.2.2.9 Quality of Life by Euro-Qol-5 |
| | Table | 14.2.2.9-1 | Frequency tables for quality of life (single dimensions) |
| | Table | 14.2.2.9-2 | Frequency tables for quality of life (dichotomized single dimensions) |
| | Table | 14.2.2.9-3 | Descriptive summary statistics for quality of life (VAS) |
| | | | 14.2.2.10 Vital signs |
| | Table | 14.2.2.10-1 | Descriptive summary statistics for vital signs |
| | Table | 14.2.2.10-2 | Frequency tables for vital signs |
| | | | 14.3 Safety analysis |
| | | | 14.3.1 Extent of exposure |

|---------------------------|----------|--------------|
| <br>WI.A.IX.C.O. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

| Table | 14.3.1-1 | Descriptive summary statistics for extent of exposure |
|---|---|---|
| | | 14.3.2 Adverse events |
| Table | 14.3.2-1 | Frequencies for adverse events |
| Table | 14.3.2-2 | Frequencies for treatment-emergent adverse events by SOC, |
| | | PT and causality |
| Listing | 14.3.2-3 | Overview of adverse events |
| Listing | 14.3.2-4 | Deaths and serious adverse events |
| | | 14.3.3 Clinical laboratory |
| Table | 14.3.3-1 | Descriptive summary statistics for laboratory values |
| Listing | 14.3.3-2 | Overview of laboratory values |
| | | 14.3.4 Vital signs |
| Table | 14.3.4-1 | Descriptive summary statistics for vital signs |
| | | 14.3.5 ECG |
| Table | 14.3.5-1 | Frequency tables for ECG overall interpretation |
| | | 14.3.6 Biomarker |
| Table | 14.3.6-1 | Descriptive summary statistics for biomarker results |
| | | 14.3.7 Other safety assessments |
| Listing | 14.3.7-1 | Echocardiography |
| Listing | 14.3.7-2 | Pregnancy test |
| Listing | 14.3.7-3 | Arterial blood collection |
| Listing | 14.3.7-4 | Assessments for APACHE II score |
| Listing | 14.3.7-5 | Assessment for evaluation of organ dysfunction (SOFA score |
| Listing | 14.3.7-6 | Daily fluid balance |
| Listing | 14.3.7-7 | Vasopressor therapy |
| | | 14.4 Pharmacokinetic data analysis |
| Table | 14.4-1 | Descriptive summary statistics for PK parameters |
| Table | 14.4-2 | Frequency tables for PK parameters |
| Listing | 14.4-3 | Individual time courses of Adrecizumab |
| Figure | 14.4-4 | Individual time courses for 2 mg/kg Adrecizumab (linear scale |
| Figure | 14.4-5 | Individual time courses for 4 mg/kg Adrecizumab (linear scale |
| Figure | 14.4-6 | Individual time courses for 2 mg/kg Adrecizumab (semi-log. scale) |
| Figure | 14.4-7 | Individual time courses for 4 mg/kg Adrecizumab (semi-log. scale) |
| Figure | 14.4-8 | Geometric means of Adrecizumab (linear scale) |
| Figure | 14.4-9 | Geometric means of Adrecizumab (semi-log. scale) |
| | | 14.5 Sensitivity analyses |
| | | 14.5.1 SSI within 14 days |
| Table | 14.5.1-1 | SSI evaluation |
| Table | 14.5.1-2 | Descriptive summary statistics for SSI within 14 days |
| Figure | 14.5.1-3 | Histogram for SSI within 14 days (Placebo vs. Adrecizumab) |
| Figure | 14.5.1-4 | Histogram for SSI within 14 days (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |

|---------------------------|----------|--------------|
| WI.7 (.1 (. O. O. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

| | | 14.5.2 Mortality |
|---|---|---|
| Figure | 14.5.2-1 | Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab) |
| Figure | 14.5.2-2 | Kaplan-Meier plot for 90-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |
| Figure | 14.5.2-3 | Kaplan-Meier plot for 28-day follow-up by treatment group (Placebo vs. Adrecizumab) |
| Figure | 14.5.2-4 | Kaplan-Meier plot for 28-day follow-up by treatment group (Placebo vs. Adrecizumab 2 mg/kg vs. Adrecizumab 4 mg/kg) |

<sup>\*</sup> will be provided in the context of topline analysis

|---------------------------|----------|--------------|
| <br>W.71.11.0.0. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

# 12. Contents of appendices

# 16 Appendices

| 16.1.9 | Documentation of statistical methods |
|---|---|
| 16.1.9-1 | Non-parametric Wilcoxon test for SSI within 14 days |
| 16.1.9-2 | Non-parametric Wilcoxon test for SSI within 28 days |
| 16.1.9-3 | Non-parametric Wilcoxon test for pSSI within 14 days |
| 16.1.9-4 | Non-parametric Wilcoxon test for pSSI within 28 days |
| 16.1.9-5 | Non-parametric Wilcoxon test for SSI cardiac component within 14 days |
| 16.1.9-6 | Non-parametric Wilcoxon test for SSI cardiac component within 28 days |
| 16.1.9-7 | Non-parametric Wilcoxon test for SSI respiratory component within 14 days |
| 16.1.9-8 | Non-parametric Wilcoxon test for SSI respiratory component within 28 days |
| 16.1.9-9 | Non-parametric Wilcoxon test for SSI renal failure component within 14 days |
| 16.1.9-10 | Non-parametric Wilcoxon test for SSI renal failure component within 28 days |
| 16.1.9-11 | Non-parametric Wilcoxon test for SSI death component within 14 days |
| 16.1.9-12 | Non-parametric Wilcoxon test for SSI death component within 28 days |
| 16.1.9-13 | Non-parametric Wilcoxon test for SSI within 14 days excl. renal component |
| 16.1.9-14 | Non-parametric Wilcoxon test for SSI within 28 days excl. renal component |
| 16.1.9-15 | Non-parametric Wilcoxon test for pSSI within 14 days excl. renal component |
| 16.1.9-16 | Non-parametric Wilcoxon test for pSSI within 28 days excl. renal component |
| 16.1.9-17 | Non-parametric Wilcoxon test for SSI within 14 days where mortality is given |
| | extra weight |
| 16.1.9-18 | Cox regression for day 28 mortality |
| 16.1.9-19 | Cox regression for day 90 mortality |

# 16.2 Patient data listings

Raw data listings will be generated and numbered appropriately.

| | MARCO | Version: | 1.0 |
|------|---------------------------|----------|--------------|
| | WI.7 (.1 (. C. C. | Date: | 05FEB2020 |
| Stat | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

# 13. Definition of Scores

# 13.1. SOFA Score

| SOFA Score | | 0 | 1 | 2 | 3 | 4 |
|---|---|---|---|---|---|---|
| Organ system | Parameter | | | | | |
| Respiratory system | PaO <sub>2</sub> / FiO <sub>2</sub> (mmHg) | ≥ 400 | < 400 | < 300 | < 200 <b>and</b><br>mechanically<br>ventilated | < 100 <b>and</b><br>mechanically<br>ventilated |
| Nervous<br>system | Glasgow<br>Coma Scale | 15 | 13 to 14 | 10 to 12 | 6 to 9 | < 6 |
| Cardiovascular<br>system | Mean arterial pressure OR administration of vasoactive agents required | No<br>hypotension | MAP < 70<br>mmHg | dopamine ≤ 5<br>μg/kg/min or<br>dobutamine<br>(any dose) | dopamine > 5<br>μg/kg/min OR<br>epinephrine ≤ 0.1<br>μg/kg/min OR<br>norepinephrine ≤ 0.1<br>μg/kg/min | dopamine > 15<br>μg/kg/min OR<br>epinephrine > 0.1<br>μg/kg/min OR<br>norepinephrine > 0.1<br>μg/kg/min |
| Liver | Bilirubin<br>(mg/dL)<br>[µmol/L] | < 1.2<br>[< 20] | 1.2 to 1.9<br>[20 to 32] | 2.0 to 5.9<br>[33 to 101] | 6.0 to 11.9<br>[102 to 204] | ≥ 12.0<br>[> 204] |
| Coagulation | Platelets<br>x10³/µl | ≥ 150 | 100 to < 150 | 50 to < 100 | 20 to < 50 | < 20 |
| Kidneys | Creatinine<br>(mg/dL)<br>[µmol/l]<br>or urine<br>output | < 1.2<br>[< 110] | 1.2 to 1.9<br>[110 to 170] | 2.0 to 3.4<br>[171 to 299] | 3.5 to 4.9<br>[300 to 440]<br>or urine output < 500<br>ml/day | ≥ 5.0<br>[> 440]<br>or urine output < 200<br>ml/day |

Template T 4.6.2-1, Version 5.0

|---------------------------|----------|--------------|
| M.71.11.C.O. | Date: | 05FEB2020 |
| Statistical Analysis Plan | Project: | ADR-02 |
| | | (AdrenOSS-2) |

# 13.2. APACHE II Score

# A. Total Acute Physiology Score (sum of points for the 12 variables below)

| | Physiologic Variable | High Abn | High Abnormal Range | | | | | Low Abnormal Range | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Filysiologic variable | +4 | +3 | +2 | +1 | 0 | +1 | +2 | +3 | +4 |
| 1 | Temperature – rectal (°C) | ≥ 41 | 39 to < 41 | | 38.5 to < 39 | 36 to < 38.5 | 34 to <<br>36 | 32 to < 34 | 30 to < 32 | <30 |
| 2 | Mean Arterial Pressure (mmHg) | > 159 | > 129 to<br>159 | > 109 to<br>129 | | > 69 to<br>109 | | > 49 to 69 | | ≤ 49 |
| 3 | Heart Rate (bpm) | ≥ 180 | 140 to < 180 | 110 to <<br>140 | | 70 to <<br>110 | | 55 to < 70 | 40 to < 55 | < 40 |
| 4 | Respiratory Rate (breaths/min) | ≥ 50 | 35 to < 50 | | 25 to < 35 | 12 to < 25 | 10 to <<br>12 | 6 to < 10 | | < 6 |
| 5 | Oxygenation: | | | | | | | | | |
| | if FiO <sub>2</sub> < 50% record PaO <sub>2</sub> | | | | | > 70 | 61 to 70 | | 55 to 60 | < 55 |
| | otherwise use A-a gradient | > 499 | 350 to 499 | 200 to 349 | | < 200 | | | | |
| 6 | Arterial pH (preferred) | ≥ 7.7 | 7.6 to < 7.7 | | 7.5 to < 7.6 | 7.33 to < 7.5 | | 7.25 to < 7.33 | 7.15 to < 7.25 | < 7.15 |
| 7 | Serum Sodium (mmol/L) | ≥ 180 | 160 to < | 155 to <<br>160 | 150 to <<br>155 | 130 to <<br>150 | | 120 to <<br>130 | 111 to <<br>120 | < 111 |
| 8 | Serum Potassium (mmol/L) | ≥ 7 | 6 to < 7 | | 5.5 to < 6 | 3.5 to < 5.5 | 3 to < 3.5 | 2.5 to < 3 | | < 2.5 |
| 9 | Serum creatinine (mg/dl) *double point score for acute renal failure | ≥ 3.5 * | 2 to < 3.5 | 1.5 to < 2 | | 0.6 to <<br>1.5 | | < 0.6 | | |
| 10 | Hematocrit (%) | ≥ 60 | | 50 to < 60 | 46 to < 50 | 30 to < 46 | | 20 to < 30 | | < 20 |
| 11 | White Blood Count (total/mm <sup>3</sup> in 1000s) | ≥ 40 | | 20 to < 40 | 15 to < 20 | 3 to < 15 | | 1 to < 3 | | < 1 |
| 12 | Glasgow Coma Scale (GCS) | | 15 – GCS Score | | | | | | | |

Template T 4.6.2-1, Version 5.0

| M.A.R.C.O. Statistical Analysis Plan | MARCO | Version: | 1.0 |
|---|---|---|---|
| | WI.71.11.C.O. | Date: | 05FEB2020 |
| | Statistical Analysis Plan | Project: | ADR-02 |
| | | | (AdrenOSS-2) |

#### B. Age points

| Age<br>(years) | Points |
|----------------|--------|
| ≤ 44 | 0 |
| 45 – 54 | 2 |
| 55 – 64 | 3 |
| 65 -74 | 5 |
| ≥ 75 | 6 |

#### C. Chronic Health Points

If the patient has a history of severe organ system insufficiency or is immunocompromised as defined below, assign points as follows:

5 points for nonoperative or emergency postoperative patients

2 points for elective postoperative patients

**Definitions:** 

The following defines "chronic organ insufficiency" and immunocompromised:

- **Liver insufficiency** biopsy proven cirrhosis, documented portal hypertension, episodes of past upper GI bleeding attributed to portal hypertension, prior episodes of hepatic failure/encephalopathy/coma
- Cardiovascular New York Heart Association Class IV Heart Failure
- Respiratory Chronic restrictive, obstructive or vascular disease resulting in severe exercise restriction (i.e., unable to climb stairs or perform household duties), documented chronic hypoxia, hypercapnia, secondary polycythemia, severe pulmonary hypertension (> 40 mmHg), respirator dependency
- Renal receiving chronic dialysis
- **Immunosuppression** the patient has received therapy that suppresses resistance to infection (e.g., immunosuppression, chemotherapy, radiation, long term or recent high dose steroids, or has a disease that is sufficiently advanced to suppress resistance to infection, e.g., leukemia, lymphoma, AIDS)

Total APACHE II Score: add together the points from A, B and C

|---------------------------|----------|--------------|
| Statistical Analysis Plan | Date: | 05FEB2020 |
| | Project: | ADR-02 |
| | | (AdrenOSS-2) |

#### 14. References

[1] Heyland et al.; Persistent organ dysfunction plus death: a novel, composite outcome measure for critical care trials. Critical Care 2011, 15

[2] https://www.mdcalc.com/sequential-organ-failure-assessment-sofa-score#next-steps (last checked 27-NOV-2019)

[3] https://www.mdcalc.com/apache-ii-score#evidence (last checked 27-NOV-2019)